CLINICAL TRIAL: NCT02928809
Title: Effect of Low-level Laser Administered to the Masseter and Anteriortemporal Muscles Prior to the Induction of Fatigue
Brief Title: Effect of Low-level Laser Prior to the Induction of Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Camila Haddad Leal de Godoy, Doctoral Student, University of Nove de Julho
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: LLLMF
Record Dates: First submitted 2016-09-30; First posted 2016-10-10 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Temporomandibular Joint Disorders
Keywords: temporomandibular joint; temporomandibular disorder; muscle fatigue; low-level laser therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TMD control (No Intervention): Patients with diagnosis of temporomandibular disorder and that are not submitted to pre-fatigue low-level laser therapy
- TMD LLL (Experimental): Patients with diagnosis of temporomandibular disorder and that are submitted to pre-fatigue low-level laser therapy
  Interventions: Device: low-level laser therapy
- Without TMD control (No Intervention): Patients without diagnosis of temporomandibular disorder and that are not submitted to pre-fatigue low-level laser therapy
- Without TMD LLL (Experimental): Patients without diagnosis of temporomandibular disorder and that are submitted to pre-fatigue low-level laser therapy
  Interventions: Device: low-level laser therapy
- TMD placebo (Placebo Comparator): Patients with diagnosis of temporomandibular disorder and that are submitted to placebo low-level laser treatment
  Interventions: Other: Placebo comparator
- Without TMD placebo (Placebo Comparator): Patients without diagnosis of temporomandibular disorder and that are submitted to placebo low-level laser treatment
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Device: low-level laser therapy — Three points will be irradiated over the masseter muscle (upper, middle and lower bundles) and one point will be irradiated over the anterior temporal muscle of each side of the face in the groups submitted to pre-fatigue laser. The following parameters will be employed: wavelength: 780 nm; energy density: 25 J/cm2; output power: 50 mW; power density: 1.25 W/cm2; and exposure time: 20 seconds per points, resulting in a total energy of 1 J per point. The laser will be applied punctually with a conventional tip in contact with the skin considering an area of 0.04 cm2.
  Arms: TMD LLL; Without TMD LLL
Other: Placebo comparator — The same equipment will be used in the placebo group, but with a pen that emits a red guide light and a warning sound, but without the emission of a laser beam.
  Arms: TMD placebo; Without TMD placebo

SUMMARY:
The objective of this study is to perform an evaluation of the effect of LLLT on the prevention of fatigue in the masseter and anterior temporal muscles in young individuals with and without TMD.

DETAILED DESCRIPTION:
Male and female individuals aged 18 to 23 years will be evaluated. The Research Diagnostic Criteria for Temporomandibular Disorders will be applied for the determination of the presence or absence of temporomandibular disorder. Each group (with and without temporomandibular disorder) will then be randomly allocated into a control group and experimental group submitted to pre-fatigue low-level laser therapy. Before and after the induction of fatigue, all volunteers will be evaluated with regard to the range of mandibular movement, bite force, sensitivity to palpation of the muscles evaluated and muscle fatigue. Low-level laser therapy will be administered to the masseter and anterior temporal muscles prior to the induction of fatigue, which will be induced with the use of chewing gum. The data will be submitted to descriptive statistical analysis. The chi-square test and Fisher's exact test will be used to establish the associations of the categorical variables. Pearson correlation coefficients will be calculated for the analysis of the correlation of the continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals aged 18 to 23 years with a signed statement of informed consent will be included in the study.

Exclusion Criteria:

* Individuals in orthodontic or orthopedic treatment for the jaws, psychological treatment or physical therapy and those who make use of muscle relaxants, anti-inflammatory agents or bite plates will be excluded from the study.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-12; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change on Bite Force | 6 minutes
  A digital dynamometer will be used for the determination of bite force. The measurements will be taken in the region of the 1st molars.

SECONDARY OUTCOMES:
Change on range of mandibular movements | 6 minutes
  The individuals will be instructed to open their mouths as wide as possible and maximum active vertical mandibular movement (distance between maxillary and mandibular central incisors) will be recorded with the aid of digital calipers. The individuals will then be instructed to repeat the motion with pressure applied to the maxillary and mandibular teeth to obtain maximum passive vertical mandibular movement with the aid of the calipers. These measurements will be made before and after LLLT.

OTHER OUTCOMES:
Change on pain upon palpation | 6 minutes
  The visual analog scale will be used before and after treatment to record pain upon palpation of the masseter and anterior temporal muscles. This is a numerical scale ranging from 0 (absence of pain) to 10 (worst pain imaginable) points.
Muscle fatigue | 6 minutes
  Muscle fatigue will be measured using the visual analog scale, which is a subjective measure that consists of a 10-centimeter line with 0 (absence of fatigue) printed at one end and 10 (maximum fatigue) printed at the other end.

CONTACTS AND LOCATIONS:
Overall Officials: Camila HL Godoy, MS, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No